CLINICAL TRIAL: NCT03725254
Title: Curative Chemoradiotherapy Versus Radical Surgery for Retroperitoneal or Paraaortic Lymph Node Recurrence of Colorectal Cancer
Brief Title: CRT Versus Surgery for Retroperitoneal or Paraaortic Lymph Node Recurrence of CRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-008
Record Dates: First submitted 2018-10-10; First posted 2018-10-31 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer; Retroperitoneal Lymph Node Metastasis; Para-aortic Lymph Node Metastasis
Keywords: Chemoradiotherapy; retroperitoneal lymphadenectomy; IMRT; SBRT
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lymph Node Excision; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radical surgery (Active Comparator): In this arm, patients with retroperitoneal or paraaortic lymph node recurrence will receive radical surgery.
  Interventions: Procedure: lymphadenectomy
- radical chemoradiotherapy (Experimental): In this arm, patients with retroperitoneal or paraaortic lymph node recurrence will receive radical chemoradiotherapy.
  Interventions: Radiation: chemoradiotherapy

INTERVENTIONS:
Procedure: lymphadenectomy — The retroperitoneal lymphadenectomy includes all lymph, fat, and connective tissue in the retroperitoneal space.
  Arms: radical surgery
Radiation: chemoradiotherapy — Radiation therapy is highly appropriate, based on the characteristics of the lesion and the surrounding critical organs, and select IMRT or stereotactic radiotherapy (SBRT).
  Arms: radical chemoradiotherapy

SUMMARY:
The study aims to compare the effects of chemoradiation versus radical surgery in treating retro-peritoneal or para-aortic lymph node metastasis in colorectal cancer. By prolonging patients' progression-free survival, local control rate and overall survival, investigators can conclude the best regimen for colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* A medical history of colorectal cancer
* Pathological or clinical diagnosis of retroperitoneal/para-vascular lymph node metastases, and located below the level of renal veins.
* The treatment target is no evidence of disease (NED), including 3 cohorts:

A. Initial treatment (primary lesion + retroperitoneal LN oligometastasis); B. Postoperative retroperitoneal/paravascular LN oligometastase; C. Postoperative retroperitoneal/paravascular LN metastasis with other organ metastases (up to NED)

* ECOG PS 0-2
* Ability to follow the program during the study period
* Signing written informed consent

Exclusion Criteria:

* Retroperitoneal LN metastasis is above the level of the renal vein.
* Unable to reach NED.
* Previous pelvic radiotherapy, the field of irradiation overlaps with this time.
* Pregnancy or breastfeeding women.
* Those with other history of malignant disease in the last 5 years, except for cured skin cancer and cervical carcinoma in situ.
* If there is an uncontrolled history of epilepsy, central nervous system disease or mental disorder, the investigator may determine that the clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
* Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention, Or a history of myocardial infarction in the last 12 months
* Organ transplantation requires immunosuppressive therapy
* Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases
* Subjects Blood routine and biochemical indicators do not meet the following criteria: hemoglobin ≥ 90g / L; absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; platelets ≥ 100 × 109 / L; ALT, AST≤2.5 times normal upper limit; ALP≤2.5 times normal upper limit; serum total bilirubin <1.5 times normal upper limit; serum creatinine <1 times normal upper limit; serum albumin ≥30g/L

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of disease progressed for any reason, assessed up to 5 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works. Also called PFS.

SECONDARY OUTCOMES:
overall survival | From date of randomization until the date of death from any cause, assessed up to 5 years
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive. In a clinical trial, measuring the overall survival is one way to see how well a new treatment works. Also called OS.
local control rate | From date of randomization until the date of disease recurrece, assessed up to 5 years
  no recurrence of the retroperitoneal or paraaortic lymph node region.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China